CLINICAL TRIAL: NCT07132970
Title: Assessment of the Leakage Rate of Ileo-colic Sutured Anastomoses Using a Polydioxanone Based Suture Material After Laparoscopic or Open Right Hemicolectomy to Treat Malignancy
Brief Title: Leakage Rate of Ileo-COlic Sutured Anastomosis After Right Hemicolectomy
Acronym: LICOSARH
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-25123
Record Dates: First submitted 2025-07-02; First posted 2025-08-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Anastomotic Leak; Colon Cancer; Right Hemicolectomy
MeSH Terms: conditions — Anastomotic Leak; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Monoplus Suture Material — Ileocolic Anastomosis Construction using Monoplus Suture Material after open or laparoscopic surgery

SUMMARY:
The primary aim of the study is to show that the ileo-colic anastomosis leakage rate until the first 30 days after surgery using MonoPlus® suture material for anastomosis construction after right hemicolectomy is not inferior to the anastomosis leakage rate published in the literature for totally handsewn or stapled-handsewn ileo-colic anastomosis.

DETAILED DESCRIPTION:
The study will include patients with right colon cancer, treated with elective colectomy and with local curative intention, in whom primary anastomosis with no protective stoma will be performed. Right colectomy is defined as a resection of terminal 10 cm of ileum, the cecum, the ascending right colon, and right third or half of the transverse colon followed by ileo-colostomy.The anastomosis leakage rate after right-sided hemicolectomy is the most important complication, because it leads to further morbidity of the affected patients. The anastomosis leakage rate ranges between 1-10% depending on the study population (cancer patients vs. non-cancer patients) and the type of anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary, elective either open or laparoscopic right hemicolectomy or right extended hemicolectomy due to malignancy with the creation of an intracorporeal or extracorporeal ileo-colic anastomosis.
* Either complete hand-sewn anastomosis or partial sutured anastomosis (e.g. combination of stapling and suturing)
* Open or laparoscopic as well as conversion from open to laparoscopic surgery
* Absence of peritoneal carcinomatosis
* Absence of vascular, nervous or bone infiltration
* Age ≥ 18 years
* Written data protection declaration (Written Informed consent)

Exclusion Criteria:

* Left hemicolectomy or left extended hemicolectomy or sigma resection
* Inflammatory bowel disease (e.g. Crohn´s disease)
* Emergency surgery
* Previous abdominal surgery with bowel resection
* Re-operation of an anastomosis (anastomosis revision surgery)
* Need for stoma creation
* Non-compliant patients
* Participation in an interventional randomized controlled study (RCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective, primary open or laparoscopic right hemicolectomy or right extended hemicolectomy for malignancy with the creation of an intracorporeal or extracorporeal ileo-colic anastomosis.
Sampling Method: Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomosis leakage | until 30 days postoperatively
  An anastomosis leak is defined as " leak of luminal contents from a anastomotic site between two hollow viscera" diagnosed (1) radiologically, by a radiographic enema with hydro soluble contrast or by computerized tomography with the presence of intra-abdominal collection adjacent to the anastomosis; (2) clinically with evidence of extravasation of bowel content or gas through a wound or drain; (3) by endoscopy, or (4) intraoperatively.
  Anastomosis leak will be classified and graded according to Clavien-Dindo.
  Grade I:
  Anastomosis leakage requiring no active intervention (e.g. antibiotics)
  Grade II:
  Anastomosis leakage requiring active radiological intervention but manageable without surgical intervention.
  Grade III:
  Anastomosis leakage requiring surgical re-intervention.
  Grade IV:
  Anastomosis leakage leading to life-threatening condition requiring IC /ICU management
  Grade V:
  Anastomosis leakage leading to death of the patient

SECONDARY OUTCOMES:
Rate of complications | discharge, 30 days postoperatively, 1 year postoperatively
  Stenosis
  * bleeding
  * hemmorage
  * obstruction
  * intradominal abszess
  * ileus
  * peritonitis
  * sepsis
Mortality rate | 30 days postoperatively, 1 year postoperatively
Surgical Site infection rate | 30 days and 12 months after surgery
  Superficial Surgical Site Infection and deep Surgical Site Infection rate according to CDC
Length of hospital stay | day of discharge after surgery
Handling of the used suture material | interoperatively
  Different dimensions rated by the surgeon using 5-point Likert scale. (1= best to 5=worse) A 5-point Likert scale is a survey tool that allows respondents to express their level of agreement or disagreement with a statement, providing nuanced feedback through five ordered response options.
  Structure of a 5-Point Likert Scale
  A typical 5-point Likert scale includes the following response options:
  Strongly Disagree: Indicates a firm rejection of the statement. Disagree: Shows a general opposition to the statement, but less intense than "Strongly Disagree." Neither Agree Nor Disagree: Represents a neutral position, suggesting indecision or a balanced view.
  Agree: Expresses support for the statement, but not with full intensity. Strongly Agree: Demonstrates strong approval or endorsement of the statement. 2
Patient satisfaction | 30 days postoperavely, 12 months postoperatively
  Assessment of patient satisfaction using 100 point scale (1 lowest- 100 highest satisfaction)
Quality of Life, using EQ5D5L | preoperatively, 30 day postoperatively and 12 months postoperatively
  EQ-5D-5L consists of 2 pages - descriptive system and the EQ visual Analogue scale (EQ-VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the respondents self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled "the best health you can imagine" and " the worst health you can imagine"
Bowel function assessment | Day of discharge after surgery, 30 days postoperatively, 1 year postoperatively
  Low Anterior Rectum Syndrome (LARS) questionnaire, assessed by the patient. The LARS Score was developed in 2012 and represents an international, validated, simple and quick instrument to assess bowel function and allows quantitative evaluation of severity of functional defects. It consists of 5 questions with a score that ranges from 0 to 42 points, with classification of patients into: no LARS (0-20), minor LARS (21-29) or major LARS (30-42 points). The five very disabling bowel symptoms of LARS score (any flatus or liquid incontinence, altered stool frequency, faecal clustering and faecal urgency) will be analysed and rated by the patients, because of their known negative influence on quality of life.
Hernia rate | 12 months postoperatively
  Hernia will be evaluated according to the EHS classification (European Hernia Society), Incisional hernia is defined as an "abdominal wall gap with or without bulge in the area of a postoperative scar perceptible or palpable by clinical examination or imaging" according to the definition to the European Hernia society

CONTACTS AND LOCATIONS:
Overall Officials: Markus Golling, Prof. Dr., Study Chair — Diak Klinikum Landkreis Schwäbisch Hall, Dept. of General Surgery
Locations (1):
- Diakonie-Klinikum Landkreis Schwäbisch Hall, Schwäbisch Hall, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No